CLINICAL TRIAL: NCT05604911
Title: Investigation of Kidney Transplant Patients for Antibodies and T-cells After Herpes Virus Vaccination and Infection
Brief Title: Herpes Virus Infections in Kidney Transplant Patients
Acronym: HINT
Status: Active, not recruiting | Type: Observational
Sponsor: Susanne Dam Nielsen, MD, DMSc (Other)
Collaborators: Technical University of Denmark (Other); Aarhus University Hospital (Other); Odense University Hospital (Other)
Responsible Party: Sponsor-Investigator, Susanne Dam Nielsen, MD, DMSc, Professor, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Other Study IDs: H-22042603; 0073947 (Other Grant/Funding Number: Novo Nordisk Foundation)
Record Dates: First submitted 2022-09-19; First posted 2022-11-03 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Kidney Transplant; Complications; Varicella Zoster Virus Infection; Vaccine-Preventable Diseases
Keywords: Varicella Zoster Virus; Shingrix; Kidney transplant; Immune response; Varicella Zoster Virus infection; Herpes Zoster; Shingles; Humane Herpes Virus 3
MeSH Terms: conditions — Varicella Zoster Virus Infection; Vaccine-Preventable Diseases; Chickenpox; Herpes Zoster

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral blood mononuclear cells (PBMC) and plasma samples will be collected and stored in a biobank.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Kidney transplant patients

SUMMARY:
Kidney transplant recipients are at increased risk of infections, including Varicella-zoster virus (VZV) infections. Vaccination against VZV is routinely offered to all kidney transplant recipients and candidates in Denmark. In this exploratory observational study, the VZV specific immune response in kidney transplant candidates and recipients will be characterized at different time points in relation to transplantation, vaccination and infections. More knowledge on the immune reaction to transplantation, VZV vaccination and VZV infections may provide improved strategies for prevention and treatment of VZV infections in kidney transplant candidates and recipients.

DETAILED DESCRIPTION:
Kidney transplantation is a life-saving procedure for patients with kidney failure, and in 2021, 252 kidney transplantations were performed in Denmark. Varicella-zoster virus (VZV) is a vaccine-preventable disease that causes varicella during primary infection and herpes zoster when reactivated later in life. VZV is one of the most common infections after organ transplantation, and kidney transplant recipients have high risk of herpes zoster (annual incidence: 3 per 100). Furthermore, kidney transplant recipients that acquire herpes zoster have high risk of disseminated and severe disease as well as increased risk of post-herpetic neuralgia.

Until 2021, the only available VZV/herpes zoster vaccines in Europe were live vaccines, and live vaccines are contraindicated in immunosuppressed individuals due to the risk of infection with the vaccine strain. However, a new, non-live, recombinant subunit herpes zoster vaccine (Shingrix®) that can be used in immunosuppressed individuals was recently approved and became available in Denmark in October 2021.

The efficacy of Shingrix® in healthy individuals is excellent (90%) both with regard to preventing herpes zoster and post-herpetic neuralgia. However, organ transplant recipients receive high doses of immunosuppressive medication, and information on efficacy and immunogenicity of Shingrix® in immunosuppressed individuals is sparse. One randomized study found the efficacy of the vaccine to be good (68%) in patients after hematopoietic stem cell transplantation. Furthermore, one phase III randomized, placebo-controlled study was conducted in 246 kidney transplant recipients, and the vaccine was found to be safe and to induce antibody responses, but the study was not powered to demonstrate efficacy.

At present, international guidelines recommend vaccination against herpes zoster prior to or after transplantation, but there is no information about the optimal timing of vaccination or duration of the immune response in transplant recipients.

Poor or no antibody response after vaccinations are documented among organ transplant recipients. Vaccination prior to transplantation or early post-transplantation may be of benefit because patients are at the highest risk of infections early post-transplantation due to high load of immunosuppressive therapy, however, this is also the period with the highest risk of non-response to vaccines. It is therefore of great importance, for both individual patients and for society, to determine the optimal timing of vaccination, response rates and duration of protection prior to use of vaccines in organ transplant recipients.

The investigators will conduct a prospective observational exploratory study including kidney transplant candidates and recipients who are offered Shingrix® vaccination. Shingrix® vaccination is routine care, and vaccination is not a part of the study, and acceptance of vaccination is not mandatory to participate in the study. The study is a national collaboration that includes all Danish kidney transplantation centers and kidney transplant recipients from all Danish regions. The study has potential to contribute with necessary information to design optimal programs for vaccine roll-out and thereby to reduce the incidence of herpes zoster and herpes zoster-related complications including hospital admissions in kidney transplant recipients as well as other solid organ transplant recipients. Furthermore, the investigators will explore differences in the immune systems of kidney transplant recipients who get VZV infections and those who don't.

The study aims to include 875 patients, of which 500 will be kidney transplant recipients (250 who are 6-12 months post-transplantation, 125 who are 12-18 months post-transplantation and 125 who are >24 months post-transplantation) and 375 kidney transplant candidates from the kidney transplant waitlist.

For participants on the transplant waitlist, blood will be collected at inclusion and 1, 2, 6 and 12 months post-inclusion, as well as 6 and 12 months post-transplantation and in the case of VZV infection. For participants who are already transplanted at inclusion, blood will be collected at inclusion, and 1, 2, 6 and 12 months post-inclusion and in the case of VZV infection. Plasma and peripheral blood mononuclear cells (PBMC) will be stored in a biobank.

All participants will be asked at inclusion to fill out a questionnaire regarding health, lifestyle, and vaccine history. At follow-ups, participants will be asked to fill out a questionnaire regarding changes in VZV infection history, vaccination history, transplant related factors and medication. Furthermore, health data will be collected from hospital records and national registries. Measurement of VZV glycoprotein E antibodies will be done using enzyme-linked immunosorbent assays (ELISA). Identification and phenotyping of VZV-specific T cells will be done through DNA-barcode labelling and flow cytometry. Cytokine profiling will be done using a Luminex MILLIPLEX assay. Analyses will be performed at the Technical University of Denmark.

ELIGIBILITY:
Inclusion Criteria:

* Kidney transplant recipient transplanted after 2019-01-01 OR on the kidney transplant waitlist
* Has been offered Shingrix® vaccination

Exclusion Criteria:

* Lack of informed consent
* Inability to understand the study information

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Kidney transplant recipients transplanted after 2019-01-01 and kidney transplant candidates followed at Copenhagen University Hospital - Rigshospitalet, Aarhus University Hospital and Odense University Hospital who has been offered Shingrix® vaccination will be invited to participate
Sampling Method: Non-Probability Sample
Enrollment: 280 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Change in levels of antibodies against Varicella-Zoster virus | 12 months
  Measurement of the change in levels of antibodies against Varicella-Zoster virus glycoprotein E using enzyme-linked immunosorbent assays (ELISA). The change will be assessed at regular intervals up to 12 months after inclusion or transplantation as well as well as in the case of infection.
Change in presence and function of Varicella-Zoster virus-specific T cells | 12 months
  Identification, phenotyping and cytokine profiling of Varicella-Zoster virus-specific T cells using DNA-barcode marking, flow cytometry and plasma cytokine profiles at regular intervals up to 12 months after inclusion or transplantation as well as in the case of infection.

CONTACTS AND LOCATIONS:
Overall Officials: Susanne D Nielsen, MD, DMSc, Principal Investigator — Department of Infectious Diseases, Copenhagen University Hospital - Rigshospitalet; Søren S Sørensen, MD, DMSc, Study Chair — Department of Nephrology, Copenhagen University Hospital - Rigshospitalet; Claus Bistrup, MD, PhD, Study Chair — Department of Nephrology, Odense University Hospital; Henrik Birn, MD, PhD, DMSc, Study Chair — Department of Nephrology, Aarhus University Hospital; Sine R Hadrup, MSc, PhD, Study Chair — Department of Health Technology, Technical University of Denmark; Annemette Hald, RN, Study Director — Department of Infectious Diseases, Copenhagen University Hospital - Rigshospitalet; Sunil K Saini, MSc, PhD, Study Director — Department of Health Technology, Technical University of Denmark; Isik S Johansen, MD, DMSc, Study Director — Department of Infectious Diseases, Odense University Hospital; Helle Bruunsgaard, MD, PhD, DMSc, Study Director — Department of Clinical Immunology, Copenhagen University Hospital - Rigshospitalet; Carsten S Larsen, MD, DMSc, Study Director — Department of Infectious Diseases, Aarhus University Hospital; Zitta B Harboe, MD, PhD, Study Director — Department of Pulmonary and Infectious Diseases, Copenhagen University Hospital - North Zealand; Moisés A Suarez Zdunek, MD, Study Director — Department of Infectious Diseases, Copenhagen University Hospital - Rigshospitalet; Sebastian R Hamm, BSc.med., Study Director — Department of Infectious Diseases, Copenhagen University Hospital - Rigshospitalet
Locations (5):
- Denmark (5):
  - Department of Nephrology, Aarhus University Hospital, Aarhus
  - Department of Infectious Diseases, Copenhagen University Hospital - Rigshospitalet, Copenhagen
  - Department of Nephrology, Copehagen University Hospital - Rigshospitalet, Copenhagen
  - Department of Health Technology, Technical University of Denmark, Lyngby
  - Department of Nephrology, Odense University Hospital, Odense

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hamm SR, Saini SK, Hald A, Vaaben AV, Pedersen NW, Suarez-Zdunek MA, Harboe ZB, Bruunsgaard H, Johansen IS, Larsen CS, Bistrup C, Birn H, Sorensen SS, Hadrup SR, Nielsen SD. Herpes Virus Infections in Kidney Transplant Patients (HINT) - a prospective observational cohort study. BMC Infect Dis. 2023 Oct 16;23(1):687. doi: 10.1186/s12879-023-08663-5. PMID 37845608